CLINICAL TRIAL: NCT03154203
Title: The Study of Non-Invasive Aortic Ambulatory Blood Pressure Monitoring for The Detection of Target Organ Damage in The Population Of Chinese Patient (SAFAR-China)
Brief Title: Non-Invasive Aortic Ambulatory Blood Pressure Monitoring for The Detection of Target Organ Damage in The Chinese Population
Acronym: SAFAR-China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director of Department of Cardiology, Professor of Tongji University, FACC, Shanghai 10th People's Hospital
Other Study IDs: SAFAR-CN
Record Dates: First submitted 2017-05-07; First posted 2017-05-16 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Blood Pressure; Cardiovascular Risk Factor; Target Organ Damage; Cardiovascular Events; Cardiovascular Mortality; Overall Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention in this study — No intervention in this study

SUMMARY:
This study is a sub-investigation of SAFAR study. Consecutive patients with established hypertension (treated or untreated with antihypertensive drugs) or with suspected hypertension are recruited and their 24-hour brachial and aortic blood pressures, cardiovascular risk factors and target organ damage are assessed. And the participants' target organ damage, cardiovascular events, cardiovascular and overall mortality will be followed four years later.

DETAILED DESCRIPTION:
SAFAR study is an ongoing perspective study which is performed in Greek. We have been participated this study and now we are going to expand this study in Chinese population.

In Shanghai Tenth People's Hospital, we recruit consecutive patients who meet the including criteria. And their medical and family history are obtained with standardized structured questionnaire including information about smoking and drinking and exercise habits, history of diabetes mellitus, cardio-cerebrovascular disease, renal disease and peripheral arterial disease, use of antihypertensive, lipid-regulating and hypoglycemic drugs. Their biochemical examinations of venous blood and urine were measured after an overnight fast.

For the 24-hour brachial and aortic ambulatory blood pressure monitoring of each patient, we use the Mobil-O-Graph NG apparatus (IEM, Stolberg, Germany), which is well validated and now commercially available.

All participants underwent carotid and cardiac ultrasonography by a validated ultrasound system (Mylab 30 CV machine, ESAOTE SPA, Genoa, Italy). The parameters of cardiac function and structure and the parameters of carotid arteries are assessed according to the ASE recommendation. Further, we use these parameters to estimate the damage of heart and carotid artery including left ventricular mass index (LVMI), carotid left ventricular diastolic function (LVDD), intima-media thickness (CIMT) and cross-sectional area(CCSA).

Four years later, the above measurements will be performed again and the corresponding data of events and mortality will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients with established hypertension (treated or untreated with antihypertensive drugs) or with suspected hypertension

Exclusion Criteria:

* Age<18 years old
* the absence of sinus rhythm during BP monitoring
* any modification in cardiovascular disease medication in the past month
* inability to provide informed consent or unwillingness/inability to adhere to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with established hypertension (treated or untreated with antihypertensive drugs) or with suspected hypertension
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 4 years
cardiovascular and all-cause mortality | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Aissopou EK, Argyris AA, Nasothimiou EG, Konstantonis GD, Tampakis K, Tentolouris N, Papathanassiou M, Theodossiadis PG, Papaioannou TG, Stehouwer CD, Sfikakis PP, Protogerou AD. Ambulatory Aortic Stiffness Is Associated With Narrow Retinal Arteriolar Caliber in Hypertensives: The SAFAR Study. Am J Hypertens. 2016 May;29(5):626-33. doi: 10.1093/ajh/hpv145. Epub 2015 Aug 24. PMID 26304958
- [Result] Zhang Y, Kollias G, Argyris AA, Papaioannou TG, Tountas C, Konstantonis GD, Achimastos A, Blacher J, Safar ME, Sfikakis PP, Protogerou AD. Association of left ventricular diastolic dysfunction with 24-h aortic ambulatory blood pressure: the SAFAR study. J Hum Hypertens. 2015 Jul;29(7):442-8. doi: 10.1038/jhh.2014.101. Epub 2014 Nov 13. PMID 25391758
- [Result] Protogerou AD, Argyris AA, Papaioannou TG, Kollias GE, Konstantonis GD, Nasothimiou E, Achimastos A, Blacher J, Safar ME, Sfikakis PP. Left-ventricular hypertrophy is associated better with 24-h aortic pressure than 24-h brachial pressure in hypertensive patients: the SAFAR study. J Hypertens. 2014 Sep;32(9):1805-14. doi: 10.1097/HJH.0000000000000263. PMID 24999798